CLINICAL TRIAL: NCT05299086
Title: As Needed Versus Regular Use of Intranasal Corticosteroid in Children With Perennial Allergic Rhinitis: A Randomized Controlled Trial
Brief Title: As Needed Versus Regular Intranasal Corticosteroid in Children With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Orathai Piboonpocanun, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 059/2565
Record Dates: First submitted 2022-03-08; First posted 2022-03-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Perennial Allergic Rhinitis; Child, Only
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Intervention Model Description: double-blinded placebo controlled randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- As needed INCs (Placebo Comparator): Use placebo everyday, and INCs as needed when the nasal symptom aggravated
  INCs = Fluticasone furoate nasal spray Placebo = Normal saline nasal spray
  Doses Fluticasone furoate nasal spray (27.5 mg/spray) age<12 yr:1 spray once daily 12 yr and older: 2 sprays once daily Normal saline nasal spray age<12 yr:1 spray once daily 12 yr and older: 2 sprays once daily
  Interventions: Drug: Intranasal Drug (INCS = Fluticasone furoate nasal spray, Placebo = Normal saline nasal spray)
- Regular INCs (Active Comparator): Use INCs everyday, and placebo as needed when the nasal symptom aggravated
  INCs = Fluticasone furoate nasal spray Placebo = Normal saline nasal spray
  Doses Fluticasone furoate nasal spray (27.5 mg/spray) age<12 yr:1 spray once daily 12 yr and older: 2 sprays once daily Normal saline nasal spray age<12 yr:1 spray once daily 12 yr and older: 2 sprays once daily
  Interventions: Drug: Intranasal Drug (INCS = Fluticasone furoate nasal spray, Placebo = Normal saline nasal spray)

INTERVENTIONS:
Drug: Intranasal Drug (INCS = Fluticasone furoate nasal spray, Placebo = Normal saline nasal spray) — The investigators want to compare the efficacy of intranasal corticosteroid between daily versus as needed use in children with perennial allergic rhinitis which had not been studied before.
  Other Names: As needed Fluticasone furoate nasal spray; Regular Fluticasone furoate nasal spray

SUMMARY:
Allergic rhinitis in children is common. According to the international study of asthma and allergies in childhood (ISAAC) phase III, the global prevalence of allergic rhinitis among children is increasing to 40.1% and the prevalence of allergic rhinitis in Bangkok area in 2018, among children aged 6-7 and 13-14 years was 16.32%. This disease is a global health problem affecting quality of life of patients in daily life, work, study and sleep.

Intranasal corticosteroid is the most effective treatment for allergic rhinitis. From real world evidence; most of allergic rhinitis patient use the drug when symptoms worsen. In children, the use of intranasal corticosteroid may cause minor local side effects such as dryness, burning sensation or epistaxis. In some intranasal corticosteroid, long-term use may result in decreased growth compared to placebo which make parents concern.

The investigators interested in studying the efficacy of intranasal corticosteroid comparing between daily use and as needed use in children with allergic rhinitis. To study the appropriate form of treatment to increase cooperation. Patient will have a better quality of life and reduce the risk of side effects from prolonged use of intranasal corticosteroid. From the literature review, it was found that most studies were conducted among adult patients with seasonal allergic rhinitis In Thailand in 2020, Thongngam et al. studied the efficacy of intranasal corticosteroid was compared between daily use and as needed use in adult patients with perennial allergic rhinitis. The results of the study concluded that the daily use group can reduced more TNSS (total nasal symptoms score) but was not statistically significant and had a greater increase in peak nasal inspiratory flow (PNIF) compared to as needed group. Interestingly, the quality of life assessment (RCQ-36 score) in both2 groups improved equally, In as needed group, the cumulative dose was 51% lower than the daily dose group.

The investigators want to compare the efficacy of intranasal corticosteroid between daily versus as needed use in children with perennial allergic rhinitis which had not been studied before.

DETAILED DESCRIPTION:
8 week Double-blinded placebo controlled randomized controlled trial to compare the efficacy between as-needed and regular use of INCS in children with perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Children patient (age 6 - 18 yr)
* Mild persistent, Moderate to severe intermittent and persistent perennial allergic rhinitis
* Rhinitis proven sensitization to aeroallergen by positive skin prick test or specific IgE result within 12 month before study recruitment
* Mean TNSS = 4 during 7 day duration before randomization (after a washout period, discontinuation of the medications listed in exclusion criteria

Exclusion Criteria:

* Patients with rhinosinusitis, nasal polyps, or significant deviated nasal septum
* Patients with a history of uncontrolled asthma, chronic lung disease, cardiovascular, hepatic, or renal diseases
* Patients taking oral or nasal decongestants within 7 d
* Patients taking INCS within 4 week
* Patients taking systemic corticosteroid within 8 week
* Patients taking H1 antihistamine within 1 week
* Patients taking antileukotriene within 4 week
* Patients who were currently or previously treated with allergen immunotherapy
* Patients with a history of upper respiratory tract infection within 14 d
* Patients with primary and secondary immune deficiency

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
TNSS (total nasal symptoms score) | 8 week
  change in TNSS 4 nose symptoms (sneezing, itching nose, watery running nose and blockage) The minimum score is 0 and maximum score is 3 each symptoms (__/12) higher scores mean worse outcome.
VAS score (Visual analog scale score for rhinitis) | 8 week
  change in VAS score Score is 0 - 10 mm higher scores mean worse outcome.

SECONDARY OUTCOMES:
Ocular symptoms score | 8 week
  Change in ocular symptoms score 2 eye symptoms (tearing eyes, itching eyes/red eyes) The minimum score is 0 and maximum score is 3 each symptoms (__/6) Higher scores mean worse outcome.
Peak nasal inspiratory flow (PNIF) | 8 week
  Change in peak nasal inspiratory flow (PNIF)
Rhinoconjunctivitis Quality of Life-36 Questionnaire score (RCQ-36) | 8 week
  Change in rhinoconjunctivitis Quality of Life-36 Questionnaire score (RCQ-36)
Medications score Medications score | 8 week
  Change in medications score Medication score Oral and/or topical (eyes or nose) non-sedative H1 antihistamines (H1A)=1 Intranasal corticosteroids (INS) with/without H1A =2 Oral corticosteroids with/without INS, with/without H1A =3 Total daily medication score (dMS) 0-3 Higher scores mean worse outcome.
Nasal FENO (nasal nitric oxide) | 8 week
  Change in nasal FENO
Nasal cytology | 8 week
  Change in nasal cytology
  Grading Nasal Cytograms A. Epithelial cells Normal morphology N Abnormal morphology A Ciliocytophthoria CCP
  B. Eosinophils, neutrophils 0* None 0 0.1-1.0* ½+ 1.1-5.0* 1+ 6.0-15.0* 2+ 16.0-20.0* 3+ >20.0* 4+
  C. Basophilic cells 0 None 0 0.1-0.3* ½+ 0.4-1.0* 1+ 1.1-3.0* 2+ 3.1-6.0* 3+ >6.0* 4+
  D. Bacteria N/A+ None 0 N/A+ 1+ N/A+ 2+ N/A+ 3+ N/A+ 4+
  E. Goblet cells# 0-24% 1+ 25-49% 2+ 50-74% 3+ 75-100% 4+
  * Mean of cells per 10 high power fields (x1000). + Note presence of intracellular bacteria. # Ratio of goblet cells to epithelial cells, expressed as percent.
Combined symptom and medication score | 8 week
  Change in combined symptom and medication score Cumulative of (nasal symptoms score + ocular symptoms score)/3 and medication score The minimum score is 0 maximum score is 6, (__/6) Higher scores mean worse outcome.
  Pfaar et al., EAACI Position Paper: 'clinical outcomes used in allergen immunotherapy trials, Allergy 69 (2014) 854-867
Correlation VAS versus TNSS, PNIF and RCQ-36 | 8 week
  VAS score (Visual analog scale score for rhinitis) total nasal symptoms score Peak nasal inspiratory flow (PNIF) Rhinoconjunctivitis Quality of Life-36 Questionnaire score (RCQ-36)
Cumulative INCs dose | 8 week
  weight the nasal spray bottles (both Fluticasone furoate nasal spray and normal saline nasal spray) on digital scale each visit and record to compare INCS used in each group

CONTACTS AND LOCATIONS:
Overall Officials: Orathai Piboonpocanun, Principal Investigator — Siriraj Hospital
Locations (1):
- Division of Allergy and Immunology, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Lunn M, Craig T. Rhinitis and sleep. Sleep Med Rev. 2011 Oct;15(5):293-9. doi: 10.1016/j.smrv.2010.12.001. Epub 2011 Feb 11. PMID 21316270
- [Background] Fokkens W, Lund V, Mullol J; European Position Paper on Rhinosinusitis and Nasal Polyps group. European position paper on rhinosinusitis and nasal polyps 2007. Rhinol Suppl. 2007;20:1-136. PMID 17844873
- [Background] Tewfik TL, Mazer B. The links between allergy and otitis media with effusion. Curr Opin Otolaryngol Head Neck Surg. 2006 Jun;14(3):187-90. doi: 10.1097/01.moo.0000193190.24849.f0. PMID 16728898
- [Background] Brozek JL, Bousquet J, Baena-Cagnani CE, Bonini S, Canonica GW, Casale TB, van Wijk RG, Ohta K, Zuberbier T, Schunemann HJ; Global Allergy and Asthma European Network; Grading of Recommendations Assessment, Development and Evaluation Working Group. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines: 2010 revision. J Allergy Clin Immunol. 2010 Sep;126(3):466-76. doi: 10.1016/j.jaci.2010.06.047. PMID 20816182
- [Background] Brozek JL, Bousquet J, Agache I, Agarwal A, Bachert C, Bosnic-Anticevich S, Brignardello-Petersen R, Canonica GW, Casale T, Chavannes NH, Correia de Sousa J, Cruz AA, Cuello-Garcia CA, Demoly P, Dykewicz M, Etxeandia-Ikobaltzeta I, Florez ID, Fokkens W, Fonseca J, Hellings PW, Klimek L, Kowalski S, Kuna P, Laisaar KT, Larenas-Linnemann DE, Lodrup Carlsen KC, Manning PJ, Meltzer E, Mullol J, Muraro A, O'Hehir R, Ohta K, Panzner P, Papadopoulos N, Park HS, Passalacqua G, Pawankar R, Price D, Riva JJ, Roldan Y, Ryan D, Sadeghirad B, Samolinski B, Schmid-Grendelmeier P, Sheikh A, Togias A, Valero A, Valiulis A, Valovirta E, Ventresca M, Wallace D, Waserman S, Wickman M, Wiercioch W, Yepes-Nunez JJ, Zhang L, Zhang Y, Zidarn M, Zuberbier T, Schunemann HJ. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines-2016 revision. J Allergy Clin Immunol. 2017 Oct;140(4):950-958. doi: 10.1016/j.jaci.2017.03.050. Epub 2017 Jun 8. PMID 28602936
- [Background] Bousquet J, Schunemann HJ, Togias A, Bachert C, Erhola M, Hellings PW, Klimek L, Pfaar O, Wallace D, Ansotegui I, Agache I, Bedbrook A, Bergmann KC, Bewick M, Bonniaud P, Bosnic-Anticevich S, Bosse I, Bouchard J, Boulet LP, Brozek J, Brusselle G, Calderon MA, Canonica WG, Caraballo L, Cardona V, Casale T, Cecchi L, Chu DK, Costa EM, Cruz AA, Czarlewski W, D'Amato G, Devillier P, Dykewicz M, Ebisawa M, Fauquert JL, Fokkens WJ, Fonseca JA, Fontaine JF, Gemicioglu B, van Wijk RG, Haahtela T, Halken S, Ierodiakonou D, Iinuma T, Ivancevich JC, Jutel M, Kaidashev I, Khaitov M, Kalayci O, Kleine Tebbe J, Kowalski ML, Kuna P, Kvedariene V, La Grutta S, Larenas-Linnemann D, Lau S, Laune D, Le L, Lieberman P, Lodrup Carlsen KC, Lourenco O, Marien G, Carreiro-Martins P, Melen E, Menditto E, Neffen H, Mercier G, Mosgues R, Mullol J, Muraro A, Namazova L, Novellino E, O'Hehir R, Okamoto Y, Ohta K, Park HS, Panzner P, Passalacqua G, Pham-Thi N, Price D, Roberts G, Roche N, Rolland C, Rosario N, Ryan D, Samolinski B, Sanchez-Borges M, Scadding GK, Shamji MH, Sheikh A, Bom AT, Toppila-Salmi S, Tsiligianni I, Valentin-Rostan M, Valiulis A, Valovirta E, Ventura MT, Walker S, Waserman S, Yorgancioglu A, Zuberbier T; Allergic Rhinitis and Its Impact on Asthma Working Group. Next-generation Allergic Rhinitis and Its Impact on Asthma (ARIA) guidelines for allergic rhinitis based on Grading of Recommendations Assessment, Development and Evaluation (GRADE) and real-world evidence. J Allergy Clin Immunol. 2020 Jan;145(1):70-80.e3. doi: 10.1016/j.jaci.2019.06.049. Epub 2019 Oct 15. PMID 31627910
- [Background] Skoner DP, Rachelefsky GS, Meltzer EO, Chervinsky P, Morris RM, Seltzer JM, Storms WW, Wood RA. Detection of growth suppression in children during treatment with intranasal beclomethasone dipropionate. Pediatrics. 2000 Feb;105(2):E23. doi: 10.1542/peds.105.2.e23. PMID 10654983
- [Background] Lee LA, Sterling R, Maspero J, Clements D, Ellsworth A, Pedersen S. Growth velocity reduced with once-daily fluticasone furoate nasal spray in prepubescent children with perennial allergic rhinitis. J Allergy Clin Immunol Pract. 2014 Jul-Aug;2(4):421-7. doi: 10.1016/j.jaip.2014.04.008. Epub 2014 May 21. PMID 25017530
- [Background] Skoner DP, Berger WE, Gawchik SM, Akbary A, Qiu C. Intranasal triamcinolone and growth velocity. Pediatrics. 2015 Feb;135(2):e348-56. doi: 10.1542/peds.2014-1641. PMID 25624374
- [Background] Juniper EF, Guyatt GH, O'Byrne PM, Viveiros M. Aqueous beclomethasone diproprionate nasal spray: regular versus "as required" use in the treatment of seasonal allergic rhinitis. J Allergy Clin Immunol. 1990 Sep;86(3 Pt 1):380-6. doi: 10.1016/s0091-6749(05)80101-0. PMID 2212409
- [Background] Juniper EF, Guyatt GH, Archer B, Ferrie PJ. Aqueous beclomethasone dipropionate in the treatment of ragweed pollen-induced rhinitis: further exploration of "as needed" use. J Allergy Clin Immunol. 1993 Jul;92(1 Pt 1):66-72. doi: 10.1016/0091-6749(93)90039-i. PMID 8335858
- [Background] Jen A, Baroody F, de Tineo M, Haney L, Blair C, Naclerio R. As-needed use of fluticasone propionate nasal spray reduces symptoms of seasonal allergic rhinitis. J Allergy Clin Immunol. 2000 Apr;105(4):732-8. doi: 10.1067/mai.2000.105225. PMID 10756223
- [Background] Kaszuba SM, Baroody FM, deTineo M, Haney L, Blair C, Naclerio RM. Superiority of an intranasal corticosteroid compared with an oral antihistamine in the as-needed treatment of seasonal allergic rhinitis. Arch Intern Med. 2001 Nov 26;161(21):2581-7. doi: 10.1001/archinte.161.21.2581. PMID 11718589
- [Background] Dykewicz MS, Kaiser HB, Nathan RA, Goode-Sellers S, Cook CK, Witham LA, Philpot EE, Rickard K. Fluticasone propionate aqueous nasal spray improves nasal symptoms of seasonal allergic rhinitis when used as needed (prn). Ann Allergy Asthma Immunol. 2003 Jul;91(1):44-8. doi: 10.1016/S1081-1206(10)62057-1. PMID 12877448
- [Background] Wartna JB, Bohnen AM, Elshout G, Pijnenburg MW, Pols DH, Gerth van Wijk RR, Bindels PJ. Symptomatic treatment of pollen-related allergic rhinoconjunctivitis in children: randomized controlled trial. Allergy. 2017 Apr;72(4):636-644. doi: 10.1111/all.13056. Epub 2016 Oct 28. PMID 27696447
- [Background] Thongngarm T, Wongsa C, Phinyo P, Assanasen P, Tantilipikorn P, Sompornrattanaphan M. As-Needed Versus Regular Use of Fluticasone Furoate Nasal Spray in Patients with Moderate to Severe, Persistent, Perennial Allergic Rhinitis: A Randomized Controlled Trial. J Allergy Clin Immunol Pract. 2021 Mar;9(3):1365-1373.e6. doi: 10.1016/j.jaip.2020.09.057. Epub 2020 Oct 10. PMID 33049392
- [Background] Bunnag C, Leurmarnkul W, Jareoncharsri P, Ungkanont K, Tunsuriyawong P, Kosrirukvongs P, Sriussadaporn P, Musiksukont S, Kosawanon S, Chairojkanjana K. Development of a health-related quality of life questionnaire for Thai patients with rhinoconjunctivitis. Asian Pac J Allergy Immunol. 2004 Jun-Sep;22(2-3):69-79. PMID 15565942
- [Background] Pfaar O, Demoly P, Gerth van Wijk R, Bonini S, Bousquet J, Canonica GW, Durham SR, Jacobsen L, Malling HJ, Mosges R, Papadopoulos NG, Rak S, Rodriguez del Rio P, Valovirta E, Wahn U, Calderon MA; European Academy of Allergy and Clinical Immunology. Recommendations for the standardization of clinical outcomes used in allergen immunotherapy trials for allergic rhinoconjunctivitis: an EAACI Position Paper. Allergy. 2014 Jul;69(7):854-67. doi: 10.1111/all.12383. Epub 2014 Apr 25. PMID 24761804
- [Background] Klimek L, Bergmann KC, Biedermann T, Bousquet J, Hellings P, Jung K, Merk H, Olze H, Schlenter W, Stock P, Ring J, Wagenmann M, Wehrmann W, Mosges R, Pfaar O. Visual analogue scales (VAS): Measuring instruments for the documentation of symptoms and therapy monitoring in cases of allergic rhinitis in everyday health care: Position Paper of the German Society of Allergology (AeDA) and the German Society of Allergy and Clinical Immunology (DGAKI), ENT Section, in collaboration with the working group on Clinical Immunology, Allergology and Environmental Medicine of the German Society of Otorhinolaryngology, Head and Neck Surgery (DGHNOKHC). Allergo J Int. 2017;26(1):16-24. doi: 10.1007/s40629-016-0006-7. Epub 2017 Jan 19. PMID 28217433
- [Background] Aneeza WH, Husain S, Rahman RA, Van Dort D, Abdullah A, Gendeh BS. Efficacy of mometasone furoate and fluticasone furoate on persistent allergic rhinoconjunctivitis. Allergy Rhinol (Providence). 2013 Fall;4(3):e120-6. doi: 10.2500/ar.2013.4.0065. PMID 24498516
- [Background] Jirapongsananuruk O, Vichyanond P. Nasal cytology in the diagnosis of allergic rhinitis in children. Ann Allergy Asthma Immunol. 1998 Feb;80(2):165-70. doi: 10.1016/S1081-1206(10)62950-X. PMID 9494449
- [Result] Bjorksten B, Clayton T, Ellwood P, Stewart A, Strachan D; ISAAC Phase III Study Group. Worldwide time trends for symptoms of rhinitis and conjunctivitis: Phase III of the International Study of Asthma and Allergies in Childhood. Pediatr Allergy Immunol. 2008 Mar;19(2):110-24. doi: 10.1111/j.1399-3038.2007.00601.x. Epub 2007 Jul 25. PMID 17651373
- [Result] Chinratanapisit S, Suratannon N, Pacharn P, Sritipsukho P, Vichyanond P. Prevalence and risk factors of allergic rhinitis in children in Bangkok area. Asian Pac J Allergy Immunol. 2019 Dec;37(4):232-239. doi: 10.12932/AP-120618-0337. PMID 30525743
- [Result] Katelaris CH, Lee BW, Potter PC, Maspero JF, Cingi C, Lopatin A, Saffer M, Xu G, Walters RD. Prevalence and diversity of allergic rhinitis in regions of the world beyond Europe and North America. Clin Exp Allergy. 2012 Feb;42(2):186-207. doi: 10.1111/j.1365-2222.2011.03891.x. Epub 2011 Nov 3. PMID 22092947